CLINICAL TRIAL: NCT04255043
Title: Intravascular Ultrasound Versus Angiography Guided Drug-coated Balloon Treatment for Denovo Lesions in High Bleeding Risk Patients: a Prospective, Multi-center, Randomized Controlled Trial
Brief Title: Intravascular Ultrasound Versus Angiography Guided Drug-coated Balloon
Acronym: ULTIMATE-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Junjie Zhang, Vice chief of the department of cardiology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20200110-02
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: All subjects will undergo 1:1 randomization to either IVUS or Angiography-guided DCB treatment for coronary denovo lesions in patients with high bleeding risk.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will remain blinded until the final study results released.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS-guided DCB (Experimental): In the IVUS guidance group, IVUS assessment will be used before procedure, post-procedure, and at the follow-up.
  Interventions: Device: IVUS guidance
- Angiography-guided DCB (Active Comparator): In the Angiography guidance group, DCB treatment will be guided by routine coronary angiography.
  Interventions: Device: Angiography guidance

INTERVENTIONS:
Device: IVUS guidance — IVUS (Boston Scientific®) guidance + DCB (Sequent® Please) treatment
  Arms: IVUS-guided DCB
Device: Angiography guidance — DCB (Sequent® Please) treatment
  Arms: Angiography-guided DCB

SUMMARY:
Drug-coated balloon (DCB) is an alternative choice for denovo lesions in coronary artery disease patients with high bleeding risk. Intravascular ultrasound (IVUS) can provide more details of coronary anatomy and stent implantation, overcoming a number of limitations of coronary angiography. However, the benefit of IVUS-guided DCB treatment has not been investigated. This study is designed to compare IVUS-guided and Angiography-guided DCB treatment for coronary denovo lesions in patients with high bleeding risk.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial that aims to enroll 260 patients with high bleeding risk.

All patients with coronary denovo lesions suitable for DCB treatment will undergo 1:1 randomization to either IVUS guidance or Angiography guidance using the Central Randomization System.

All subjects will be screened according to the predefined inclusion and exclusion criteria per protocol. Data and images will be collected during the index procedure, and at the predefined 7-month coronary angiography follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. De novo lesions, suitable for DCB treatment.
2. Patients with high bleeding risk.

Exclusion Criteria:

1. Target lesion length > 15mm.
2. Severe calcified lesions.
3. Left main disease.
4. Ostial lesions.
5. Three-vessel disease.
6. Acute myocardial infarction within 48 hours.
7. Target vessel received stent implantation.
8. Hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
late lumen loss (LLL) at 7 months after procedure | 7 months
  LLL is defined as the difference between postprocedural minimal lumen diameter (MLD) minus MLD at the time of angiographic follow-up

SECONDARY OUTCOMES:
Target vessel failure (TVF) at 6 months | 6 months
  TVF is defined as the composite of cardiac death, target-vessel myocardial infarction and ischemia-driven target-vessel revascularization.
bleeding at 6 months | 6 months
  bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao XF, Ge Z, Kong XQ, Chen X, Han L, Qian XS, Zuo GF, Wang ZM, Wang J, Song JX, Lin L, Pan T, Ye F, Wang Y, Zhang JJ, Chen SL; ULTIMATE Ⅲ Investigators. Intravascular Ultrasound vs Angiography-Guided Drug-Coated Balloon Angioplasty: The ULTIMATE Ⅲ Trial. JACC Cardiovasc Interv. 2024 Jul 8;17(13):1519-1528. doi: 10.1016/j.jcin.2024.04.014. Epub 2024 Jun 5. PMID 38842991